CLINICAL TRIAL: NCT01592422
Title: Maintenance Immunotherapy With Autologous Cytokine-induced Killer Cells for Small Cell Lung Cancer
Brief Title: Maintenance Therapy With Autologous Cytokine-induced Killer Cells for Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Guosheng Feng, Professor, People's Hospital of Guangxi Zhuang Autonomous Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIKSCLC-2012
Record Dates: First submitted 2012-04-26; First posted 2012-05-07 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; Maintenance therapy; Immunotherapy; Autologous cytokine-induced killer cell
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunotherapy (Experimental): Subjects receive autologous cytokine-induced killer cell infusion every month
  Interventions: Biological: Autologous cytokine-induced killer cell
- Best Supportive Care (Active Comparator): Best Supportive Care
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Biological: Autologous cytokine-induced killer cell — Subjects receive autologous cytokine-induced killer cell infusion every month in the absence of disease progression or unacceptable toxicity.
  Arms: Immunotherapy
Other: Best Supportive Care — Best Supportive Care in the absence of disease progression
  Arms: Best Supportive Care

SUMMARY:
The role of maintenance therapy in the management of Small Cell Lung Cancer (SCLC) has not been confirmed. Many treatment modalities like chemotherapy, interferons and other biological agents have been tested as maintenance therapy in SCLC, but the results are disappointing. A marginal survival advantage is seen in maintenance with chemotherapy and interferon-alpha, however, the functioning status and immune system may get worse, which subsequently has a negative impact on patient's quality-of-life. Immunotherapy with autologous cytokine-induced killer (CIK) cells can activate the antitumor defense mechanism through stimulating immune response and altering the interaction between tumor and its host. This effect may result in improved tumor control and survival, as well as a better quality of life. To test the hypothesis, a randomized controlled study was conducted to compare CIK cells with best supportive care as maintenance therapy for SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven small cell lung cancer
* Patients currently receiving 4-6 cycles of chemotherapy regimen with VP-16 and a platinum-based drug as first-line therapy in the absence of disease progression
* Age between 18-75
* Performance status ≤2
* No uncontrolled metabolic disease, infection, and neurological disorders
* No congestive heart failure, severe arrhythmia, and coronal atherosclerosis heart disease
* Life expectancy more than three months.
* Without contraindication of immunotherapy with autologous cytokine-induced killer cells
* No other malignancies
* Signed study-specific consent form prior to study entry

Exclusion Criteria:

* Patients receiving other anti-tumor therapy (like thermotherapy)
* Pregnant or lactating women
* Allergy or unacceptable toxicity of immunotherapy with autologous cytokine-induced killer cells
* Uncontrolled mental disorder
* Patient having acute hepatitis virus infection, active tuberculosis, or other acute infectious diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | One year

SECONDARY OUTCOMES:
Overall survival | Two years
Quality-of-life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guosheng Feng, MD, Study Chair — People's Hospital of Guangxi Zhuang Autonomous Region; Yuan Liang, MD, Study Chair — Guangxi Department of Public Health; Hui Lin, MD, Phd, Study Chair — People's Hospital of Guangxi Zhuang Autonomous Region; Heming Lu, MD, Study Chair — People's Hospital of Guangxi Zhuang Autonomous Region
Locations (1):
- The people's Hospital of the Guangxi Zhuang Autonomous Region, Nanning, Guangxi, China